CLINICAL TRIAL: NCT05259735
Title: A Clinical Guideline-based Management of Type-2 Diabetes by Ayurvedic Practitioners in Nepal: a Feasibility Cluster Randomised Controlled Trial
Brief Title: A Clinical Guideline-based Management of Type-2 Diabetes by Ayurvedic Practitioners in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nepal Health Research Council (Other Government)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Dr. Pradip Gyanwali,MD, Executive Chief, Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayurveda DM Study
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetes; Type2Diabetes; Diabetes Mellitus
Keywords: Ayurveda; DiabetesMellitus; ClinicalGuideline
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Final outcome assessment will be conducted after 6 month for both arms by blind assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Clinical guideline-based management of T2DM by Ayurvedic practitioners. The clinical guideline will cover topics like diagnostic criteria, blood glucose targets, lifestyle advice, Ayurvedic medicines, monitoring and follow-up (including screening for complications and referral to specialists for complications management). The clinical guideline will make recommendations based on the best available evidence. Ayurvedic practitioners will have at least a 5½ year undergraduate medical degree in Ayurveda. Regular training will be provided to Ayurvedic practitioners (in groups) in the use of clinical guideline which will involve roleplaying and structured and instructive feedback to improve their performance. The trainings will be recorded on the Training Attendance Log and they will be provided a Training Certificate for completing the training.
  Interventions: Combination Product: Clinical Guideline based Management
- Comparator (Active Comparator): Comparator: Currently, no standard clinical guideline is used by Ayurvedic practitioners to manage T2DM in Nepal. Thus, the comparator will be the usual management of T2DM (i.e., without any clinical guideline) by Ayurvedic practitioners.
  Participants will continue their medications for other systemic diseases, if any.
  Interventions: Other: Comparator

INTERVENTIONS:
Combination Product: Clinical Guideline based Management — Clinical guidline based management will be done for Type 2 diabetes Mellitus
  Arms: Intervention
Other: Comparator — In this arm usual management of T2DM without any clinical guideline
  Arms: Comparator

SUMMARY:
T2DM is a complex disorder which has major health, social and economic consequences. Its chronic hyperglycaemia is associated with macro- and micro-vascular complications and even death. The prevalence of T2DM in Nepal is high.

In Nepal, Ayurveda is the dominant traditional medical system and is in use for thousands of years, especially for meeting the primary healthcare needs. Lack of availability of western medical system doctors in rural areas is another reason. In recognition of these facts, the Nepalese government actively promotes Ayurveda and deploys Ayurvedic practitioners in PHCs, often as the main clinical provider.

This is a two-arm, feasibility cluster RCT with blinded outcome assessment and integrated qualitative process evaluation will be conducted in 12 Ayurvedic Primary Health Care Center Participants who are aged 18 years or above, new T2DM patients (i.e., treatment naïve), diagnosed by the participating Ayurvedic practitioner and able to provide written informed consent will be enrolled in the study. Each participant will be involved in the study for six months.

Patient will be assessed for Glycated haemoglobin, Lipid Profile, Physiological parameters like heart rate and pulse rate, Anthropometric parameters, EuroQol-5D-5L

DETAILED DESCRIPTION:
In Nepal, Ayurveda is the dominant traditional medical system and is in use for thousands of years, especially for meeting the primary healthcare needs. The classical texts are written in Sanskrit, an ancient language. T2DM is one of the top diseases for which patients consult Ayurvedic practitioners, and many T2DM patients use Ayurvedic treatments, often from the beginning and exclusively and throughout their lives.Ayurveda fits their health beliefs and culture. Acceptability, satisfaction and perceived relief are usually high, especially among rural, poor, older and tribal populations. Many T2DM patients prefer not to use western medicines - to avoid the associated side-effects and costs and the mode of administration like insulin injections. Lack of availability of western medical system doctors in rural areas is another reason. In recognition of these facts, the Nepalese government actively promotes Ayurveda and deploys Ayurvedic practitioners in PHCs, often as the main clinical provider.

Strong concerns remain about the sub-optimal T2DM management of many patients, arising from the unacceptable variations in Ayurvedic clinical practice. The actions to be taken at different stages of the T2DM care pathway are largely left to the judgment of the individual Ayurvedic practitioner (including screening for complications and referral to specialists), resulting in these unacceptable variations. Despite the clinical effectiveness and safety of several Ayurvedic medicines for managing T2DM found in trial settings, many non-evidence based herbal and herbo-mineral medicines are prescribed by them in real practice, which can have serious adverse effects on patients, including heavy metal poisoning. It is exceedingly difficult for them to be versed with the latest data on most effective and safe Ayurvedic medicines. One of the major challenges identified by them in their clinical decision-making process and delivering quality care to T2DM patients is the absence of a good quality clinical guideline. Its absence forces many of them to blindly follow the claims made by others or use a 'trial and error' approach.

Faced with similar issues in the western medical system, clinical guidelines have been effectively deployed in every aspect of clinical care in the last few decades. For example, clinical trials conducted in English and Mexican primary care settings found that the introduction of clinical guidelines was effective in managing T2DM. Despite their pervasive use in the western medical system, their existence in Ayurvedic clinical practice remains extremely limited. Many stakeholders, including Ayurvedic practitioners, patient groups, the Nepalese government and WHO, are advocating for good quality clinical guidelines for Ayurvedic practitioners. Thus, a good quality clinical guideline, based on the best available evidence, to manage T2DM by Ayurvedic practitioners may address the problems mentioned above. We searched a range of trial registries and databases, and no study is investigating the utility of such an intervention for managing T2DM by Ayurvedic practitioners. Thus, there is a need for a robustly designed pragmatic study to evaluate such an innovative approach.

This is a two-arm, feasibility cluster RCT with blinded outcome assessment and integrated qualitative process evaluation.

12 Primary Health Centres (PHCs) with at least one Ayurvedic practitioner (most have only one) for the duration of the study and willing to participate in the study will be randomised (1:1) to intervention or comparator groups by an independent statistician according to a computer-generated randomisation schedule. PHCs should be screened for eligibility (PHC Screening and Randomisation Form) and recorded on the Screening of PHCs Eligible PHCs will be randomised and provided Site ID.

Ayurvedic practitioners and patients cannot be 'blinded' to group allocation, but the outcome assessor will be 'blind'.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* new T2DM patients (i.e., treatment naïve), diagnosed by the participating Ayurvedic practitioner
* able to provide written informed consent.

Exclusion Criteria:

* Pregnant women
* those with any serious or uncontrolled medical condition (e.g., cancer)
* those currently receiving (or has plans to receive during the study period) any related non-pharmaceutical/pharmaceutical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
To assess the change in the management of type-2 Diabetes with the introduction of Clinical Guideline | Assessment will be done from the data of screening until the 6 months
  The assessment will be done in the baseline and the end line by measuring HbA1C
To assess the change Health related quality of life with the introduction of clinical guideline | Assessment will be done from the data of screening until the 6 months
  Health related quality of life will be assessed in the baseline and the end line through HRQOL questionnaire

SECONDARY OUTCOMES:
To determine the rate of dropout | From the date of screening until the 6 months
  To compare the rate of dropout in the intervention and control group ,
To determine the number of participants who adhere to the guideline | From the date of screening until the 6 months
  To determine the rate of participants adhering to the guideline

CONTACTS AND LOCATIONS:
Overall Officials: Kaushik Chattopadhyay, MPH, Principal Investigator — University of Nottingham; Pradip Gyanwali, MD, Principal Investigator — Nepal Health Research Council
Locations (1):
- Nepal Health Research Council, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No